CLINICAL TRIAL: NCT03167749
Title: Effect of Type and Severity of Liver Cirrhosis on Semen Parameters and Reproductive Hormones
Brief Title: Effect of Liver Cirrhosis on Semen Parameters and Reproductive Hormones
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Allam, Principal investigator, Assiut University
Other Study IDs: LcRh
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: Male patients with liver cirrhosis of any etiology and severity. Laboratory tests will be done
  Interventions: Diagnostic Test: Laboratory test
- Control group: Healthy males without history or features of liver disease. Laboratory tests will be done
  Interventions: Diagnostic Test: Laboratory test

INTERVENTIONS:
Diagnostic Test: Laboratory test — Semen analysis and reproductive hormonal assay (free and total testosterone, luteinizing hormone, follicle-stimulating hormone , estradiol and prolactin hormone) for both patients and control group

SUMMARY:
Normal testicular hormonal and spermatogenic function depends not only on the testis itself, but also on the integrity of the hypothalamus and anterior pituitary. Systemic diseases has been shown to influence male gonadal function in variety of ways, leading to reduced libido, erectile impotence, infertility, osteoporosis, and decreased physical stamina and muscle mass. The effect of systemic diseases may occur directly at the testicular level: reduced Leydig cell function will lead to androgen deficiency, while diseases affecting Spermatogenesis may lead to infertility. Alternatively, acute and chronic illness may interfere with the hypothalamic-pituitary axis and lead to reduced testicular function.

DETAILED DESCRIPTION:
Liver is thoroughly involved in proteins, cytokines and interleukins synthesis and destruction. Therefore, abnormal function of endocrine organs is expected in patients with liver cirrhosis.

Hypogonadism is a frequent clinical feature in patients with liver cirrhosis. These patients have gynecomastia, decreased libido, signs of feminization, testicular atrophy and low testosterone level, as well as reduced Spermatogenesis. These features are more severe in patients with higher Child Pugh score.

Several hormonal abnormalities are responsible for these clinical alterations. Estrogen/androgen ratio has been increased in cirrhosis while there is reduction in serum testosterone and dehydroepiandrosterone level.

Hyperprolactinemia is present in patients with cirrhosis and may involve in Hypogonadism by an inhibitory effect on gonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* male patient with liver cirrhosis of any etiology and severity.

Exclusion Criteria:

1. Systemic conditions like:chronic renal failure, diabetes mellitus, thyrotoxicosis, hypothyroidism, Cushing's disease and cancer.
2. Local conditions like :Varicocele, urogenital infections, history of cryptorchidism, functional and obstructive azoospermia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: male patients with liver cirrhosis will be recruited from the department of gastroenterology and tropical medicine and other group of healthy males without history or features of liver disease serves as the control group will be recruited from the outpatient clinics at Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Semen parameters (volume, total sperm count and sperm concentration, motility and morphology) | Baseline
  Mean difference in semen parameters(volume, total sperm count and sperm concentration, motility and morphology) between patients and control group
Serum level of reproductive hormones (free and total testosterone, luteinizing hormone , follicle-stimulating hormone, estradiol and prolactin hormone) | Baseline
  Mean difference in serum level of reproductive hormones(free and total testosterone, luteinizing hormone, follicle-stimulating hormone , estradiol and prolactin hormone) between patients and control group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner HE, Wass JA. Gonadal function in men with chronic illness. Clin Endocrinol (Oxf). 1997 Oct;47(4):379-403. doi: 10.1046/j.1365-2265.1997.2611108.x. No abstract available. PMID 9404435
- [Background] Eshraghian A, Taghavi SA. Systematic review: endocrine abnormalities in patients with liver cirrhosis. Arch Iran Med. 2014 Oct;17(10):713-21. PMID 25305772
- [Background] Karagiannis A, Harsoulis F. Gonadal dysfunction in systemic diseases. Eur J Endocrinol. 2005 Apr;152(4):501-13. doi: 10.1530/eje.1.01886. PMID 15817904
- [Background] van Thiel DH, Gavaler JS, Spero JA, Egler KM, Wright C, Sanghvi AT, Hasiba U, Lewis JH. Patterns of hypothalamic-pituitary-gonadal dysfunction in men with liver disease due to differing etiologies. Hepatology. 1981 Jan-Feb;1(1):39-46. doi: 10.1002/hep.1840010107. PMID 6793494
- [Background] Bannister P, Oakes J, Sheridan P, Losowsky MS. Sex hormone changes in chronic liver disease: a matched study of alcoholic versus non-alcoholic liver disease. Q J Med. 1987 Apr;63(240):305-13. PMID 2960998
- [Background] Simon-Holtorf J, Monig H, Klomp HJ, Reinecke-Luthge A, Folsch UR, Kloehn S. Expression and distribution of prolactin receptor in normal, fibrotic, and cirrhotic human liver. Exp Clin Endocrinol Diabetes. 2006 Nov;114(10):584-9. doi: 10.1055/s-2006-948310. PMID 17177141